CLINICAL TRIAL: NCT00966251
Title: Phase I/II Safety and Tolerability Study of the Monoclonal Antibody CT-011 in Patients With Hepatocellular Carcinoma
Brief Title: Safety and Tolerability Study of the Monoclonal Antibody CT-011 in Patients With Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped because of slow accrual
Sponsor: CureTech Ltd (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-2009-02
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: Primary Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT-011 (Experimental)
  Interventions: Drug: CT-011

INTERVENTIONS:
Drug: CT-011 — CT-011

SUMMARY:
The objective of this pilot study is to evaluate the safety, tolerability and activity of the monoclonal antibody CT-011 administered intravenously to patients with Primary Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years and above, both genders.
2. Histologically or cytologically confirmed Primary Hepatocellular Carcinoma (HCC)
3. No fibrolamellar subtype HCC
4. Not eligible for any other systemic anti-neoplastic treatment approved for HCC
5. Not eligible for Transarterial chemoembolization (TACE ).
6. No more than 1 prior systemic therapy. Previous TACE or Radiofrequency ablation (RFA) that were used for HCC, are permitted.
7. Not a candidate for curative surgical resection or liver transplantation
8. Measurable disease defined by the identification at least 1 measurable lesion by MRI using RECIST criteria. Tumor in area of TACE or RFA must be enlarging post-procedure to be considered measurable disease.
9. Alpha-fetoprotein (AFP) greater than the upper limit of normal (ULN)
10. Child's Pugh classification A
11. ECOG performance status 0-1

Exclusion Criteria:

1. Patients progressing to liver failure.
2. No core biopsy within the past 7 days
3. Patients who are eligible for Transarterial Chemoembolization (TACE)
4. Patients on concurrent anti-neoplastic therapy (including interferon)
5. Patients who have received any systemic anti-neoplastic therapy not approved for the treatment of HCC.
6. Patients on concurrent steroids, other than those allowed for routine antiemetics, or inhaled steroids
7. Presence of metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of CT-011 in patients with Primary Hepatocellular Carcinoma | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel